CLINICAL TRIAL: NCT04638933
Title: Effect of CPAP Therapy on Molecular Breath Patterns in Patients With OSA (BrOSA)
Brief Title: Effect of CPAP Therapy on Molecular Breath Patterns in Patients With OSA
Acronym: BrOSA
Status: Completed | Type: Observational
Sponsor: Malcolm Kohler (Other)
Responsible Party: Sponsor-Investigator, Malcolm Kohler, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: BASEC-Nr. 2020-02084
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Exhaled breath analysis; Mass spectrometry
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSA patients: Patients with proven OSA (apnea-hypopnea index ≥20/h, ESS >10, age ≥18 years) and initiation of CPAP treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Determination of changes in molecular breath patterns in OSA patients, naïve for OSA treatment before and after one month of CPAP therapy by untargeted, secondary electrospray ionisation-high resolution mass spectrometry (SESI-HRMS). Furthermore, breath patterns will be assessed for correlation and association to clinical outcomes such as change in OSA severity, sleepiness, and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed OSA (AHI ≥20/h)
* Patient is willing to start CPAP therapy
* ESS > 10 points
* 18 years or above

Exclusion Criteria:

* Moribund or severe disease prohibiting protocol adherence
* Use of oxygen therapy or home ventilation
* Physical or intellectual impairment precluding informed consent or protocol adherence
* Known malignancy, acute pulmonary disease, drug or alcohol abuse, known active inflammatory diseases (e.g. autoimmune disease), relevant congenital defects e.g. amino acid metabolism defect, relevant endocrinological disease, renal failure (GFR < 15 mL/min)
* Pregnant patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with proven OSA (apnea-hypopnea index ≥20/h, ESS >10, age ≥18 years) and initiation of CPAP treatment
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Exhaled breath pattern | twice during 1 month
  Change in exhaled breath pattern in response to one month of CPAP treatment

SECONDARY OUTCOMES:
OSA severity parameter | twice during 1 month
  Correlation of breath print with changes in OSA severity parameters on CPAP (e.g. AHI, ODI)
Vital signs | twice during 1 month
  Correlation of breath print with changes in blood pressure and heart rate
Sleepiness | twice during 1 month
  Correlation of breath print with changes in sleepiness (Epworth sleepiness scale) and Functional outcome of sleep questionnaire (FOSQ 30)
Spirometry | twice during 1 month
  Correlation of breath print with spirometry (FEV1, FVC)
CPAP therapy | twice during 1 month
  Correlation of breath print with CPAP therapy parameters (adherence and leakage)
Therapy feedback | twice during 1 month
  Correlation of breath print with patients' and their partners' feedback report on CPAP machine used

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland